CLINICAL TRIAL: NCT02178462
Title: Evaluation of AminoIndex™ (Amino Metabolomic) As Biomarkers for Gynecologic Cancer in the U. S. Population
Brief Title: Biomarkers for Gynecologic Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ajinomoto Co., Inc. (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Other Study IDs: AI-2014-1
Record Dates: First submitted 2014-06-23; First posted 2014-06-30 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Benign Gynecological Disease
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Subject blood samples (plasma and serum) will be collected for testing at a single visit
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Primary ovarian cancer patients: Intervention will not be administered.
- Primary endometrial cancer patients: Intervention will not be administered.
- Benign gynecological disease patients: Intervention will not be administered.
- Healthy controls: Intervention will not be administered.

SUMMARY:
A novel blood metabolic biomarker, AminoIndexTM (gynecological), was developed for gynecological cancers from over 400 Japanese patient's plasma free amino acid profiles (PFAAs) by a rapid and sensitive LC-MS (Liquid Chromatography - Mass Spectrometry), followed by multivariate statistical analyses. However, further studies to assess whether this biomarker demonstrates the same performance characteristics in non-Japanese populations for cancer is yet to be determined.

DETAILED DESCRIPTION:
"AminoIndex Technology" was developed based on high-throughput and absolute quantitative analysis method of amino acids and amines using UFLC-MS, and creating a clinical database to search for amino acid patterns across different diseases including cancer. "AminoIndex Technology" can evaluate certain health conditions and the possibility of diseases by analyzing the balance of plasma amino acids. Multicenter studies in Japan were conducted to develop an blood based biomarker panel for cancer.

This study wil be conducted to evaluate the performance of AminoIndexTM (gynecological) biomarker based on "AminoIndex Technology" for gynecological cancers in US populations. This will be done by analyzing plasma metabolites including amino acids, from endometrial and ovarian cancer patients, from patients with benign gynecological disease, and healthy subjects using Liquid Chromatography and Mass Spectrometry (LC-MS) and Liquid Chromatography - Tandem Mass Spectrometry (LC-MSMS).

ELIGIBILITY:
Inclusion Criteria:

Participants in this study will be patients with Primary endometrial and ovarian cancer, benign gynecological diseases (such as uterine fibroids, endometriosis, dysplasia, and benign ovarian tumors), and healthy subjects that meet the following criteria:

* Age > 20 years (no data is currently available on use of AminoIndexTM in patients under 20 years of age or over 80 years of age)
* Willing to follow fasting and clinic visit requirements
* Ability to understand and consent to participate in study.

Women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

Women will be excluded from study participation for the following reasons:

* An inability to fast (no food or drink other than water) for 8 hours prior to the pre-surgery sample collection.
* Are known to be positive for HIV/HCV/HBV
* Pregnancy or breastfeeding (Pregnant and breastfeeding women are excluded from this study because amino acid levels are known to differ in pregnancy).
* Currently receiving investigational agents.
* History of any drug therapy or surgery for treatment of gynecological cancer
* Unable to come for the blood sample collection between 6:00 AM and 12:00 Noon
* Currently undergoing dialysis
* Congenital metabolic disease
* The investigator considers individual to be ineligible based on prior medical history, histology or other findings

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants in this study will be patients with Primary endometrial and ovarian cancer, benign gynecological diseases (such as uterine fibroids, endometriosis, dysplasia, and benign ovarian tumors), and healthy subjects that meet the following eligibility criteria:
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2014-06; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Performance characteristics of AminoIndexTM biomarker to discriminate gynecologic cancer from benign disease or healthy subjects | Baseline
  Performance characteristics of the AminoIndexTM biomarker will be evaluated by analyzing blood and comparing results between cancer patients, benign gynecological diseases, and healthy subjects. (AUC of the ROC curve, sensitivity, specificity, and other measures of performance)

SECONDARY OUTCOMES:
To identify and quantify new blood amino metabolic biomarkers that are associated with gynecologic cancer | Baseline
  Blood will be examined for new blood amino metabolic biomarkers and their concentrations will be compared between cancer patients and benign disease patients and healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: David O'Malley, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States